CLINICAL TRIAL: NCT03354429
Title: A Randomised, Double-Blind, Placebo-Controlled, International, Multicentre, Phase III Study to Investigate the Efficacy and Safety of Ticagrelor and ASA Compared With ASA in the Prevention of Stroke and Death in Patients With Acute Ischaemic Stroke or Transient Ischaemic Attack
Brief Title: THALES - Acute STroke or Transient IscHaemic Attack Treated With TicAgreLor and ASA for PrEvention of Stroke and Death
Acronym: THALES
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D5134C00003; 2016-004232-37 (EudraCT Number)
Record Dates: First submitted 2017-11-20; First posted 2017-11-28 (Actual); Results first posted 2020-12-22 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Acute Ischaemic Stroke; Transient Ischaemic Attack
Keywords: Acute ischaemic stroke; Transient Ischaemic Attack (TIA); Stroke
MeSH Terms: conditions — Ischemic Attack, Transient; Stroke | interventions — Ticagrelor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TICAGRELOR (Experimental)
  Interventions: Drug: Ticagrelor
- TICAGRELOR PLACEBO (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ticagrelor — Ticagrelor arm: Day 1, loading dose of ticagrelor followed by daily maintenance dose until Day 30.
  Arms: TICAGRELOR
Drug: Placebo — Placebo arm: Day 1, loading dose of placebo followed by placebo daily maintenance dose until Day 30.
  Arms: TICAGRELOR PLACEBO

SUMMARY:
Study to investigate if the study drug ticagrelor and ASA is more effective than Placebo (inactive tablet) and ASA in preventing new stroke events

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed informed consent prior to any study-specific procedure
2. ≥40 years of age
3. Acute onset of cerebral ischaemia due to

   1. AIS with NIHSS ≤5. AIS is defined as acute onset of neurological deficit attributed to focal brain ischaemia, and either of the following:

      * Persistent signs or symptoms of the ischaemic event at the time o randomisation, OR
      * Acute ischaemic brain lesion documented before randomisation by computed tomography (CT) scan or magnetic resonance imaging (MRI) (diffusion-weighted imaging) and that could account for the clinical presentation
   2. High-risk TIA, defined as neurological deficit of acute onset attributed to focal ischaemia of the brain by history or examination with complete resolution of the deficit, and at least one of the following:

      * ABCD2 score ≥6 and TIA symptoms not limited to isolated numbness, isolated visual changes, or isolated dizziness/vertigo
      * Symptomatic intracranial arterial occlusive disease that could account for the clinical presentation, documented by transcranial Doppler or vascular imaging and defined as at least 50% narrowing in the diameter of the vessel lumen
      * Internal carotid arterial occlusive disease that could account for the clinical presentation, documented by Doppler, ultrasound, or vascular imaging and defined as at least 50% narrowing in diameter of the vessel lumen
4. Randomisation occurring within 24 hours after onset of symptoms; for wake-up strokes (when the time of symptom onset is not known), within 24 hours from the time point at which the patient was reported to be in their normal condition
5. CT or MRI performed after symptom onset ruling out intracranial haemorrhage or other pathology, such as vascular malformation, tumour, or abscess that according

to the Investigator could explain symptoms or contraindicate study treatment

Exclusion Criteria:

1. Need for or an anticipated need for any of the following:

   1. Dual antiplatelet therapy with ASA and P2Y12 inhibitors (including patients with carotid artery stenting and percutaneous coronary intervention)
   2. Antiplatelets other than ASA (eg, GPIIb/IIIa inhibitors, clopidogrel, ticlopidine, prasugrel, dipyridamole, ozagrel, cilostazol, ticagrelor) and other antithrombotic agents with antiplatelet effects, including traditional/herbal medicine agents
   3. Anticoagulants (eg, warfarin, oral thrombin and factor Xa inhibitors, bivalirudin, hirudin, argatroban, fondaparinux, or unfractionated heparin and long-term treatment with low-molecular weight heparins). Short-term treatment (≤7 days) with low-dose low-molecular weight heparin may be used in immobilised patients at the discretion of the Investigator
2. Any history of atrial fibrillation/flutter, ventricular aneurysm, or suspicion of other cardioembolic pathology for TIA or stroke
3. Patients who should receive or have received any intravenous or intra-arterial thrombolysis or mechanical thrombectomy within 24 hours prior to randomisation
4. Planned carotid endarterectomy that requires halting investigational product within 3 days of randomisation or is expected to require unblinding of investigational product (planned carotid endarterectomy is in itself not an exclusion criterion)
5. History of previous intracranial haemorrhage at any time (asymptomatic microbleeds do not qualify), gastrointestinal haemorrhage within the past 6 months, or major surgery within 30 days
6. Patients considered to be at risk of bradycardic events (eg, known sick sinus syndrome or second- or third-degree atrioventricular block) unless already treated with a permanent pacemaker
7. Inability of the patient to understand and/or comply with study procedures and/or follow-up, in the opinion of the Investigator
8. Known hypersensitivity to ticagrelor or ASA
9. Need for or an anticipated need for oral or intravenous therapy with any of the following:

   1. Strong cytochrome P450 3A (CYP3A4) inhibitors (eg, ketoconazole, clarithromycin [but not erythromycin or azithromycin], nefazadone, ritonavir, atazanavir) that cannot be stopped for the course of the study
   2. Long-term (>7 days) non-steroidal anti-inflammatory drugs
10. Known bleeding diathesis or coagulation disorder (eg, thrombotic thrombocytopenic purpura)
11. Known severe liver disease (eg, ascites or signs of coagulopathy)
12. Renal failure requiring dialysis
13. Pregnancy or breastfeeding. Women of child-bearing potential who are not willing to use a medically accepted method of contraception that is considered reliable in the judgment of the Investigator
14. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site)
15. Previous enrolment or randomisation in the present study
16. Participation in another clinical study with an investigational product at any time during the 30 days prior to randomisation (regardless of when treatment with the investigational product was discontinued)

Ages: 40 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11016 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2019-12-13 (Actual); Study Completion 2019-12-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (295):
- Argentina (9):
  - Research Site, Adrogué
  - Research Site, Buenos Aires
  - Research Site, Capital Federal
  - Research Site, Ciudad Autónoma de Bs. As.
  - Research Site, Córdoba
  - Research Site, Mar del Plata
  - Research Site, Mendoza
  - Research Site, Rosario
  - Research Site, Salta
- Australia (6):
  - Research Site, Adelaide
  - Research Site, Heidelberg
  - Research Site, Herston
  - Research Site, Parkville
  - Research Site, Southport
  - Research Site, St Albans
- Belgium (13):
  - Research Site, Antwerp
  - Research Site, Assebroek (Brugge)
  - Research Site, Bruges
  - Research Site, Brussels
  - Research Site, Dendermonde
  - Research Site, Edegem
  - Research Site, Kortrijk
  - Research Site, Leuven
  - Research Site, Liège
  - Research Site, Ostend
  - Research Site, Roeselare
  - Research Site, Sint-Truiden
  - Research Site, Yvoir
- Brazil (9):
  - Research Site, Botucatu
  - Research Site, Curitiba
  - Research Site, Goiânia
  - Research Site, Joinville
  - Research Site, Maringá
  - Research Site, Porto Alegre
  - Research Site, Ribeirão Preto
  - Research Site, Rio de Janeiro
  - Research Site, Salvador
- Bulgaria (8):
  - Research Site, Dupnitsa
  - Research Site, Kozloduy
  - Research Site, Lukovit
  - Research Site, Pazardzhik
  - Research Site, Pleven
  - Research Site, Sliven
  - Research Site, Sofia
  - Research Site, Teteven
- Canada (4):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Lethbridge, Alberta
  - Research Site, Chicoutimi
- China (31):
  - Research Site, Baoji
  - Research Site, Baotou
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Chifeng
  - Research Site, Daqing
  - Research Site, Foshan
  - Research Site, Guangzhou
  - Research Site, Guiyang
  - Research Site, Haikou
  - Research Site, Hangzhou
  - Research Site, Hohhot
  - Research Site, Jinan
  - Research Site, Jinzhou
  - Research Site, Liuchow
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Nantong
  - Research Site, Ningbo
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Taiyuan
  - Research Site, Tangshan
  - Research Site, Tianjin
  - Research Site, Wenzhou
  - Research Site, Wuhan
  - Research Site, Wuxi
  - Research Site, Xi'an
  - Research Site, Xiamen
  - Research Site, Xining
  - Research Site, Xuzhou
- Czechia (6):
  - Research Site, Brno
  - Research Site, Chomutov
  - Research Site, Ostrava
  - Research Site, Pardubice
  - Research Site, Prague
  - Research Site, Ústí nad Labem
- France (22):
  - Research Site, Bayonne
  - Research Site, Besançon
  - Research Site, Bordeaux
  - Research Site, Bourg-en-Bresse
  - Research Site, Brest
  - Research Site, Caen
  - Research Site, Corbeil-Essonnes
  - Research Site, Dijon
  - Research Site, Le Chesnay
  - Research Site, Lille
  - Research Site, Metz
  - Research Site, Montpellier
  - Research Site, Nancy
  - Research Site, Nice
  - Research Site, Paris
  - Research Site, Rennes
  - Research Site, Rouen
  - Research Site, Saint-Herblain
  - Research Site, Saint-Priez En Jarez
  - Research Site, Strasbourg
  - Research Site, Suresnes
  - Research Site, Toulouse
- Germany (9):
  - Research Site, Altenburg
  - Research Site, Bad Neustadt an der Saale
  - Research Site, Berlin
  - Research Site, Erlangen
  - Research Site, Essen
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Minden
  - Research Site, Münster
- Hong Kong (2):
  - Research Site, Hong Kong
  - Research Site, Kowloon
- Hungary (12):
  - Research Site, Baja
  - Research Site, Balassagyarmat
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Győr
  - Research Site, Kistarcsa
  - Research Site, Miskolc
  - Research Site, Nyíregyháza
  - Research Site, Pécs
  - Research Site, Sopron-Balf
  - Research Site, Székesfehérvár
  - Research Site, Tatabánya
- India (14):
  - Research Site, Bangalore
  - Research Site, Bengaluru
  - Research Site, Dehradun
  - Research Site, Guntur
  - Research Site, Gūrgaon
  - Research Site, Hyderabad
  - Research Site, Kanpur
  - Research Site, Kolkata
  - Research Site, Mangalore
  - Research Site, Nagpur
  - Research Site, Nashik
  - Research Site, New Delhi
  - Research Site, Srikakulam
  - Research Site, Varanasi
- Italy (16):
  - Research Site, Cona
  - Research Site, Genova
  - Research Site, Massa
  - Research Site, Milan
  - Research Site, Modena
  - Research Site, Negrar
  - Research Site, Pavia
  - Research Site, Perugia
  - Research Site, Pietra Ligure
  - Research Site, Pisa
  - Research Site, Roma
  - Research Site, Siena
  - Research Site, Varese
  - Research Site, Verona
  - Research Site, Vicenza
  - Research Site, Vizzolo Predabissi
- Mexico (8):
  - Research Site, Culiacán
  - Research Site, D.F
  - Research Site, Durango
  - Research Site, Guadalajara
  - Research Site, Mexico City
  - Research Site, México
  - Research Site, Monterrey
  - Research Site, Tijuana
- Peru (5):
  - Research Site, Bellavista
  - Research Site, Callao
  - Research Site, Lima
  - Research Site, Trujillo
  - Research Site, Urb. El Chipe
- Poland (19):
  - Research Site, Bialystok
  - Research Site, Chełm
  - Research Site, Działdowo
  - Research Site, Gdansk
  - Research Site, Gmina Końskie
  - Research Site, Gmina Świebodzin
  - Research Site, Grodzisk Mazowiecki
  - Research Site, Gryfice
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Olsztyn
  - Research Site, Ostrołęka
  - Research Site, Rybnik
  - Research Site, Sandomierz
  - Research Site, Skarżysko-Kamienna
  - Research Site, Warsaw
  - Research Site, Zielona Góra
- Romania (6):
  - Research Site, Bucharest
  - Research Site, Iași
  - Research Site, Oradea
  - Research Site, Sibiu
  - Research Site, Târgu Mureş
  - Research Site, Timișoara
- Russia (17):
  - Research Site, Chelyabinsk
  - Research Site, Izhevsk
  - Research Site, Kazan'
  - Research Site, Kemerovo
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Novosibirsk
  - Research Site, Ryazan
  - Research Site, Saint Petersburg
  - Research Site, Samara
  - Research Site, Saratov
  - Research Site, Sochi
  - Research Site, Tomsk
  - Research Site, Ufa
  - Research Site, Voronezh
  - Research Site, Yaroslavl
  - Research Site, Yekaterinburg
- Saudi Arabia (2):
  - Research Site, Jeddah
  - Research Site, Riyadh
- Slovakia (11):
  - Research Site, Dolný Kubín
  - Research Site, Levoča
  - Research Site, Liptovský Mikuláš
  - Research Site, Martin
  - Research Site, Nitra
  - Research Site, Rimavská Sobota
  - Research Site, Skalica
  - Research Site, Spišská Nová Ves
  - Research Site, Trenčín
  - Research Site, Trnava
  - Research Site, Žiar nad Hronom
- South Korea (11):
  - Research Site, Anyang-si
  - Research Site, Busan
  - Research Site, Cheongju-si
  - Research Site, Daegu
  - Research Site, Daejeon
  - Research Site, Goyang-si
  - Research Site, Gwangju
  - Research Site, Incheon
  - Research Site, Jeju-do
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Spain (11):
  - Research Site, Albacete
  - Research Site, Alicante
  - Research Site, Badalona(Barcelona)
  - Research Site, Barcelona
  - Research Site, Girona
  - Research Site, Lleida
  - Research Site, Madrid
  - Research Site, Seville
  - Research Site, Valencia
  - Research Site, Valladolid
  - Research Site, Zaragoza
- Sweden (9):
  - Research Site, Gothenburg
  - Research Site, Linköping
  - Research Site, Lund
  - Research Site, Malmo
  - Research Site, Östersund
  - Research Site, Skövde
  - Research Site, Solna
  - Research Site, Stockholm
  - Research Site, Uppsala
- Taiwan (8):
  - Research Site, Changhua
  - Research Site, Kaohsiung City
  - Research Site, Keelung
  - Research Site, New Taipei City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan Hsien
- Thailand (12):
  - Research Site, Bangkok
  - Research Site, Chon Buri
  - Research Site, Hat Yai
  - Research Site, Khlong Luang
  - Research Site, Khon Kaen
  - Research Site, Lampang
  - Research Site, Muang
  - Research Site, Nakhonpathom
  - Research Site, Prachinburi
  - Research Site, Rajthevi
  - Research Site, Ratchaburi
  - Research Site, Ubonratchathani
- Ukraine (11):
  - Research Site, Chernivtsі
  - Research Site, Ivano-Frankivsk
  - Research Site, Kharkiv Region
  - Research Site, Kherson
  - Research Site, Kyiv
  - Research Site, Lutsk
  - Research Site, Lviv
  - Research Site, Poltava
  - Research Site, Ternopil
  - Research Site, Vinnytsia
  - Research Site, Zaporizhzhia
- Vietnam (4):
  - Research Site, Hanoi
  - Research Site, Hà Nội
  - Research Site, Ho Chi Minh City
  - Research Site, Đông Nãi

REFERENCES:
- [Derived] Tank A, Johnston SC, Jain R, Amarenco P, Mellstrom C, Rikner K, Denison H, Ladenvall P, Knutsson M, Himmelmann A, Evans SR, James S, Molina CA, Wang Y, Ouwens M. Cost-effectiveness of ticagrelor plus aspirin versus aspirin in acute ischaemic stroke or transient ischaemic attack: an economic evaluation of the THALES trial. BMJ Neurol Open. 2023 Aug 24;5(2):e000478. doi: 10.1136/bmjno-2023-000478. eCollection 2023. PMID 37637218
- [Derived] Johnston SC, Amarenco P, Aunes M, Denison H, Evans SR, Himmelmann A, Jahreskog M, James S, Knutsson M, Ladenvall P, Molina CA, Nylander S, Rother J, Wang Y; THALES Investigators. Ischemic Benefit and Hemorrhage Risk of Ticagrelor-Aspirin Versus Aspirin in Patients With Acute Ischemic Stroke or Transient Ischemic Attack. Stroke. 2021 Nov;52(11):3482-3489. doi: 10.1161/STROKEAHA.121.035555. Epub 2021 Sep 3. PMID 34477459
- [Derived] Wang Y, Pan Y, Li H, Amarenco P, Denison H, Evans SR, Himmelmann A, James S, Birve F, Ladenvall P, Molina CA, Johnston SC; THALES Steering Committee and Investigators. Efficacy and Safety of Ticagrelor and Aspirin in Patients With Moderate Ischemic Stroke: An Exploratory Analysis of the THALES Randomized Clinical Trial. JAMA Neurol. 2021 Sep 1;78(9):1091-1098. doi: 10.1001/jamaneurol.2021.2440. PMID 34244703
- [Derived] Yaghi S, de Havenon A, Rostanski S, Kvernland A, Mac Grory B, Furie KL, Kim AS, Easton JD, Johnston SC, Henninger N. Carotid Stenosis and Recurrent Ischemic Stroke: A Post-Hoc Analysis of the POINT Trial. Stroke. 2021 Jul;52(7):2414-2417. doi: 10.1161/STROKEAHA.121.034089. Epub 2021 May 4. PMID 33940954
- [Derived] Amarenco P, Denison H, Evans SR, Himmelmann A, James S, Knutsson M, Ladenvall P, Molina CA, Wang Y, Johnston SC; THALES Steering Committee and Investigators*. Ticagrelor Added to Aspirin in Acute Nonsevere Ischemic Stroke or Transient Ischemic Attack of Atherosclerotic Origin. Stroke. 2020 Dec;51(12):3504-3513. doi: 10.1161/STROKEAHA.120.032239. Epub 2020 Nov 16. PMID 33198608
- [Derived] Amarenco P, Denison H, Evans SR, Himmelmann A, James S, Knutsson M, Ladenvall P, Molina CA, Wang Y, Johnston SC; THALES Steering Committee and Investigators. Ticagrelor Added to Aspirin in Acute Ischemic Stroke or Transient Ischemic Attack in Prevention of Disabling Stroke: A Randomized Clinical Trial. JAMA Neurol. 2020 Nov 7;78(2):1-9. doi: 10.1001/jamaneurol.2020.4396. Online ahead of print. PMID 33159526
- [Derived] Johnston SC, Amarenco P, Denison H, Evans SR, Himmelmann A, James S, Knutsson M, Ladenvall P, Molina CA, Wang Y; THALES Investigators. Ticagrelor and Aspirin or Aspirin Alone in Acute Ischemic Stroke or TIA. N Engl J Med. 2020 Jul 16;383(3):207-217. doi: 10.1056/NEJMoa1916870. PMID 32668111
- [Derived] Johnston SC, Amarenco P, Denison H, Evans SR, Himmelmann A, James S, Knutsson M, Ladenvall P, Molina CA, Wang Y; THALES Investigators. The Acute Stroke or Transient Ischemic Attack Treated with Ticagrelor and Aspirin for Prevention of Stroke and Death (THALES) trial: Rationale and design. Int J Stroke. 2019 Oct;14(7):745-751. doi: 10.1177/1747493019830307. Epub 2019 Feb 12. PMID 30747613
- [Derived] Wong KSL, Amarenco P, Albers GW, Denison H, Easton JD, Evans SR, Held P, Himmelmann A, Kasner SE, Knutsson M, Ladenvall P, Minematsu K, Molina CA, Wang Y, Johnston SC; SOCRATES Steering Committee and Investigators. Efficacy and Safety of Ticagrelor in Relation to Aspirin Use Within the Week Before Randomization in the SOCRATES Trial. Stroke. 2018 Jul;49(7):1678-1685. doi: 10.1161/STROKEAHA.118.020553. Epub 2018 Jun 18. PMID 29915123
- See also: redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5134C00003&attachmentIdentifier=3c773278-ed11-4f6a-ba36-6d927f39a776&fileName=d5134c00003_SAP_redacted.pdf&versionIdentifier=
- See also: redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5134C00003&attachmentIdentifier=52098dc2-641a-49a8-8478-d745f5a10a26&fileName=d5134c00003_CSP_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 414 study sites in 28 countries enrolled patients. The first patient was enrolled on 22 January 2018. The last patient visit took place on 13 December 2019.
Pre-assignment Details: 11073 patients screened; 11016 patients randomised. 57 patients who were not randomised (patient did not meet inclusion/exclusion criteria n=52, patient decision n=5).
Groups:
- TICAGRELOR: Ticagrelor 180 mg day 1, followed by 90 mg twice daily day 2-30
- PLACEBO: Placebo 180 mg day 1, followed by 90 mg twice daily day 2-30
Period: Overall Study
Arm/Group | TICAGRELOR | PLACEBO
Started | 5523 | 5493
Completed | 5514 | 5486
Not Completed | 9 | 7
Not completed — Withdrawal by Subject | 8 | 7
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set including all randomised patients
Groups:
- Total: Total of all reporting groups
Arm/Group | TICAGRELOR | PLACEBO | Total
Number analyzed (Participants) | 5523 | 5493 | 11016
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.2 (11.0) | 65.1 (11.1) | 65.1 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2108 | 2171 | 4279
  Male | 3415 | 3322 | 6737
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 2973 | 2948 | 5921
  Black or African American | 21 | 32 | 53
  Asian | 2353 | 2339 | 4692
  Native Hawaiian or other Pacific Islander | 1 | 3 | 4
  American Indian or Alaska Native | 173 | 168 | 341
  Other | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Composite of Subsequent Stroke or Death
Description: Participants with subsequent stroke or death
Time Frame: From randomisation (day 1) to visit 3 (day 30-34)
Population: Full analysis set including all randomised patients
Measure: Count of Participants; unit: Participants
Arm/Group | TICAGRELOR | PLACEBO
Number analyzed (Participants) | 5523 | 5493
Participants | 303 | 362
Statistical Analysis 1: Comparison: TICAGRELOR vs PLACEBO; Test type: Superiority; p = 0.015, Regression, Cox — The hypothesis was tested at the 4.996% two-sided significance level to account for the planned interim analysis with the overall type I error preserved at 5%. A hierarchical test sequence was used to address the issue of multiple testing; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.71 to 0.96] — Placebo is the reference group (denominator)

2. Secondary Outcome: Ischaemic Stroke
Description: Number of participants with ischaemic stroke
Time Frame: From randomisation (day 1) to visit 3 (day 30-34)
Population: Full analysis set including all randomised patients
Measure: Count of Participants; unit: Participants
Arm/Group | TICAGRELOR | PLACEBO
Number analyzed (Participants) | 5523 | 5493
Participants | 276 | 345
Statistical Analysis 1: Comparison: TICAGRELOR vs PLACEBO; Test type: Superiority; p = 0.004, Regression, Cox — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.68 to 0.93] — Placebo is the reference group (denominator)

3. Secondary Outcome: Number of Participants With Modified Rankin Scale (mRS) Score >1 at Visit 3
Description: The modified Rankin Scale (mRS) is a scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. The scale runs from 0-6, running from perfect health without symptoms to death.0 - No symptoms,1 - No significant disability. Able to carry out all usual activities, despite some symptoms. 2 - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities. 3 - Moderate disability. Requires some help, but able to walk unassisted. 4 - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted. 5 - Severe disability. Requires constant nursing care and attention, bedridden, incontinent. 6 - Dead.
Time Frame: Visit 3 (day 30-34)
Population: Full analysis set including all randomised patients. Patients with missing mRS score or missing covariates, NIHSS (National Institutes of Health Stroke Scale) score and history of stroke (yes/no), were excluded
Measure: Count of Participants; unit: Participants
Arm/Group | TICAGRELOR | PLACEBO
Number analyzed (Participants) | 5386 | 5333
Participants | 1282 | 1284
Statistical Analysis 1: Comparison: TICAGRELOR vs PLACEBO; Test type: Superiority; p = 0.613, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; NIHSS (National Institutes of Health Stroke Scale) score and history of stroke (yes/no) included as covariates; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.89 to 1.07] — Placebo is the reference group (denominator)

4. Other Pre Specified Outcome: Bleeding Event That Fulfils Serious Adverse Event Criteria and is Categorised as GUSTO Severe
Description: Participants with bleeding event that fulfils serious adverse event criteria and is categorised as GUSTO Severe. GUSTO is a bleeding scale (GUSTO = Global Utilization of Streptokinase and Tissue plasminogen activator for Occluded coronary arteries). GUSTO Severe bleeding is defined as any of the following: (1) fatal bleeding, (2) intracranial bleeding, or (3) bleeding that caused haemodynamic compromise requiring intervention
Time Frame: From randomisation (day 1) to visit 3 (day 30-34)
Population: Full analysis set including all randomised patients
Measure: Count of Participants; unit: Participants
Arm/Group | TICAGRELOR | PLACEBO
Number analyzed (Participants) | 5523 | 5493
Participants | 28 | 7
Statistical Analysis 1: Comparison: TICAGRELOR vs PLACEBO; Test type: Other; p = 0.001, Regression, Cox; Hazard Ratio (HR) = 3.99, 95% CI 2-sided [1.74 to 9.14] — Placebo is the reference group (denominator)

5. Other Pre Specified Outcome: ICH or Fatal Bleeding Event
Description: Participants with ICH or fatal bleeding event
Time Frame: From randomisation (day 1) to visit 3 (day 30-34)
Population: Full analysis set including all randomised patients
Measure: Count of Participants; unit: Participants
Arm/Group | TICAGRELOR | PLACEBO
Number analyzed (Participants) | 5523 | 5493
Participants | 22 | 6
Statistical Analysis 1: Comparison: TICAGRELOR vs PLACEBO; Test type: Other; p = 0.005, Regression, Cox; Hazard Ratio (HR) = 3.66, 95% CI 2-sided [1.48 to 9.02] — Placebo is the reference group (denominator)

6. Other Pre Specified Outcome: Bleeding Event That Fulfils Serious Adverse Event Criteria and is Categorised as GUSTO Moderate/Severe
Description: Participants with bleeding event that fulfils serious adverse event criteria and is categorised as GUSTO Moderate/Severe. GUSTO is a bleeding scale (GUSTO = Global Utilization of Streptokinase and Tissue plasminogen activator for Occluded coronary arteries). GUSTO Severe bleeding is defined as any of the following: (1) fatal bleeding, (2) intracranial bleeding, or (3) bleeding that caused haemodynamic compromise requiring intervention. GUSTO Moderate bleeding is a bleeding requiring transfusion of whole blood or packed red blood cells without haemodynamic compromise
Time Frame: From randomisation (day 1) to visit 3 (day 30-34)
Population: Full analysis set including all randomised patients
Measure: Count of Participants; unit: Participants
Arm/Group | TICAGRELOR | PLACEBO
Number analyzed (Participants) | 5523 | 5493
Participants | 36 | 11
Statistical Analysis 1: Comparison: TICAGRELOR vs PLACEBO; Test type: Other; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 3.27, 95% CI 2-sided [1.67 to 6.43] — Placebo is the reference group (denominator)

7. Other Pre Specified Outcome: Premature Permanent Discontinuation of IP Due to Bleeding
Description: Participants with premature permanent discontinuation of IP due to bleeding
Time Frame: From randomisation (day 1) to visit 3 (day 30-34)
Population: Full analysis set including all randomised patients
Measure: Count of Participants; unit: Participants
Arm/Group | TICAGRELOR | PLACEBO
Number analyzed (Participants) | 5523 | 5493
Participants | 152 | 32
Statistical Analysis 1: Comparison: TICAGRELOR vs PLACEBO; Test type: Other; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 4.80, 95% CI 2-sided [3.28 to 7.02] — Placebo is the reference group (denominator)

ADVERSE EVENTS:
Time Frame: From randomisation (day 1) to visit 3 (day 30-34)
Description: Only serious adverse events (SAEs) and premature permanent discontinuations of study drug due to AEs (DAEs) were to be collected
Arm/Group | Ticagrelor | Placebo
All-Cause Mortality (participants affected / at risk) | 40/5523 | 32/5493
Serious Adverse Events (participants affected / at risk) | 571/5523 | 609/5493
Other Adverse Events (participants affected / at risk) | 0/5523 | 0/5493
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ticagrelor (N=5523) | Placebo (N=5493)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Polycythaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Spontaneous haematoma (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 4 (4) | 5 (5)
Angina unstable (Cardiac disorders) | 2 (2) | 0 (0)
Aortic valve disease mixed (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 18 (18) | 15 (17)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Atrial thrombosis (Cardiac disorders) | 4 (4) | 2 (2)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 2 (2)
Atrioventricular block second degree (Cardiac disorders) | 3 (3) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 2 (2)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac asthma (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 3 (3) | 0 (0)
Cardiac ventricular thrombosis (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 2 (2)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Congestive cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 2 (2) | 2 (2)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1)
Intracardiac thrombus (Cardiac disorders) | 2 (2) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve disease mixed (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 2 (2)
Right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Sinoatrial block (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Atrial septal defect (Congenital, familial and genetic disorders) | 1 (1) | 4 (4)
Vascular malformation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 2 (2) | 2 (2)
Vestibular ataxia (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Angle closure glaucoma (Eye disorders) | 0 (0) | 1 (1)
Diabetic retinopathy (Eye disorders) | 1 (1) | 0 (0)
Idiopathic orbital inflammation (Eye disorders) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastric disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 6 (6) | 6 (6)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3) | 0 (0)
Melaena (Gastrointestinal disorders) | 2 (2) | 0 (0)
Oesophageal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 3 (3) | 2 (2)
Rectal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 (5) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 4 (4) | 4 (4)
Device related thrombosis (General disorders) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Necrosis (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 1 (1)
Sudden cardiac death (General disorders) | 0 (0) | 1 (1)
Acute hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 2 (2)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatocellular injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 2 (2)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Brain abscess (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 3 (3)
Clostridium colitis (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 2 (2) | 0 (0)
Escherichia sepsis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal bacterial infection (Infections and infestations) | 1 (1) | 2 (2)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 0 (0)
Intervertebral discitis (Infections and infestations) | 0 (0) | 1 (1)
Klebsiella sepsis (Infections and infestations) | 0 (0) | 1 (1)
Neurosyphilis (Infections and infestations) | 1 (1) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 25 (25) | 28 (29)
Pseudomembranous colitis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis chronic (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 3 (3) | 5 (5)
Septic shock (Infections and infestations) | 2 (2) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Tracheobronchitis (Infections and infestations) | 1 (1) | 0 (0)
Tuberculosis (Infections and infestations) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 6 (6) | 7 (7)
Urinary tract infection enterococcal (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 1 (1)
Arterial bypass occlusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Open globe injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Periprocedural myocardial infarction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0)
Occult blood positive (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Sympathetic posterior cervical syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cardiac myxoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Focal nodular hyperplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Malignant mediastinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myeloproliferative neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Phaeochromocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Autonomic neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Balance disorder (Nervous system disorders) | 2 (2) | 0 (0)
Basal ganglia haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 3 (3) | 3 (3)
Brain stem stroke (Nervous system disorders) | 1 (1) | 0 (0)
Brain stem syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Carotid arteriosclerosis (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery occlusion (Nervous system disorders) | 0 (0) | 2 (2)
Carotid artery stenosis (Nervous system disorders) | 8 (8) | 7 (7)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Central pain syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cerebellar infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral artery stenosis (Nervous system disorders) | 2 (2) | 2 (2)
Cerebral haemorrhage (Nervous system disorders) | 4 (4) | 3 (3)
Cerebral infarction (Nervous system disorders) | 6 (6) | 8 (8)
Cerebral ischaemia (Nervous system disorders) | 2 (2) | 0 (0)
Cerebral venous sinus thrombosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral venous thrombosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 6 (6) | 7 (7)
Cerebrovascular disorder (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular insufficiency (Nervous system disorders) | 1 (1) | 0 (0)
Chronic inflammatory demyelinating polyradiculoneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Dementia alzheimer's type (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 3 (3)
Dysgraphia (Nervous system disorders) | 0 (0) | 1 (1)
Dysmetria (Nervous system disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 5 (5) | 3 (3)
Guillain-barre syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 2 (2) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 7 (7) | 0 (0)
Haemorrhagic transformation stroke (Nervous system disorders) | 8 (8) | 6 (6)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hemianaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 1 (1)
Hypoglycaemic seizure (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 1 (1) | 2 (2)
Ischaemic cerebral infarction (Nervous system disorders) | 4 (4) | 6 (6)
Ischaemic stroke (Nervous system disorders) | 254 (258) | 324 (330)
Lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0)
Lacunar stroke (Nervous system disorders) | 0 (0) | 2 (2)
Loss of consciousness (Nervous system disorders) | 2 (2) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Neurological symptom (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Paresis (Nervous system disorders) | 0 (0) | 1 (1)
Parkinson's disease (Nervous system disorders) | 0 (0) | 1 (1)
Partial seizures (Nervous system disorders) | 2 (2) | 0 (0)
Post stroke seizure (Nervous system disorders) | 0 (0) | 1 (1)
Psychomotor hyperactivity (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 4 (4) | 3 (3)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Spondylitic myelopathy (Nervous system disorders) | 1 (1) | 0 (0)
Status epilepticus (Nervous system disorders) | 2 (2) | 0 (0)
Stroke in evolution (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0)
Thalamic infarction (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 12 (12) | 30 (31)
Vascular dementia (Nervous system disorders) | 1 (1) | 0 (0)
Vertebral artery stenosis (Nervous system disorders) | 2 (2) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 2 (2)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 2 (2) | 0 (0)
Conversion disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 3 (3)
Hallucination, visual (Psychiatric disorders) | 1 (1) | 0 (0)
Neuropsychiatric symptoms (Psychiatric disorders) | 1 (1) | 0 (0)
Organic brain syndrome (Psychiatric disorders) | 0 (0) | 2 (2)
Panic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 2 (2) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Somatic symptom disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 4 (4) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 2 (2) | 1 (1)
Cystitis haemorrhagic (Renal and urinary disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
End stage renal disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 8 (8) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephropathy toxic (Renal and urinary disorders) | 1 (1) | 1 (1)
Prerenal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 3 (3)
Renal injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary bladder polyp (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1)
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 5 (5)
Pulmonary granuloma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Aortic dissection (Vascular disorders) | 1 (1) | 0 (0)
Aortic intramural haematoma (Vascular disorders) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1)
Arterial stenosis (Vascular disorders) | 1 (1) | 0 (0)
Arteritis (Vascular disorders) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 2 (2)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 5 (5) | 5 (6)
Hypertensive crisis (Vascular disorders) | 3 (3) | 4 (4)
Hypertensive urgency (Vascular disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Penetrating aortic ulcer (Vascular disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 2 (2)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Subclavian artery stenosis (Vascular disorders) | 0 (0) | 1 (1)
Vasculitis (Vascular disorders) | 1 (1) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-12-09): https://cdn.clinicaltrials.gov/large-docs/29/NCT03354429/SAP_000.pdf
  • Study Protocol (2019-05-08): https://cdn.clinicaltrials.gov/large-docs/29/NCT03354429/Prot_001.pdf